CLINICAL TRIAL: NCT03499977
Title: The Effects of Acute Cycling on Executive Control
Brief Title: Acute Cycling on Executive Control
Acronym: ACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Dr. Harry Prapavessis, Principal Investigator, Western University, Canada
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PA and Executive Functioning
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Physical Activity
Keywords: Physical Activity; Executive function; Anti-saccade
MeSH Terms: conditions — Motor Activity | interventions — Sitting Position

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sitting (Experimental): The participant will be asked to sit for 10 min (not increasing their heart rate) then do the anti-saccade task
  Interventions: Behavioral: Sitting
- Low-Intensity Cycling (Experimental): Participant will be asked to cycle for 10 min (<40% VO2R) and then perform the anti-saccade task
  Interventions: Behavioral: Light-Intensity Cycling
- Moderate-Intensity Cycling (Experimental): The participant will be asked to do 10 min of cycling (40-59% VO2R) followed but the anti-saccade task
  Interventions: Behavioral: Moderate-Intensity Cycling
- High-Intensity Cycling (Experimental): The participant will be asked to do 10 min of cycling (60%-84% VO2R) followed but the anti-saccade task
  Interventions: Behavioral: High-Intensity Cycling

INTERVENTIONS:
Behavioral: Sitting — 10 min bouts
  Arms: Sitting
Behavioral: Light-Intensity Cycling — 10min bout
  Arms: Low-Intensity Cycling
Behavioral: Moderate-Intensity Cycling — 10 min bout
  Arms: Moderate-Intensity Cycling
Behavioral: High-Intensity Cycling — 10 min bout
  Arms: High-Intensity Cycling

SUMMARY:
This study will examine whether 10-minute bouts of cycling at various intensities will impact executive functioning (i.e., cognitive ability) as assessed by the antisaccade (AS) task through a total of five visits. An antisaccade is a rapid eye movement away from a visual target. The ability to suppress making an eye movement towards a visual target gauges inhibitory control (i.e., a domain of executive functioning). In the initial visit, participants' exercise capacity will be assessed through a maximal effort cycling test. Intensities for the cycling bouts (i.e., high, moderate, low) in subsequent sessions will be based upon this maximal effort cycling test. In visits 2 through 5, participants will complete an AS task, followed by a 10-minute bout of cycling, and then complete the AS task again. The order of cycling intensities will be randomized between participants. Differences in the AS task (i.e., reaction time and accuracy) will be compared between and within cycling conditions.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, write and understand English
* Full time student enrolled at Western University
* Able to perform a ten-minute exercise task at a light intensity without health implications
* Have email or phone number for contacting purposes

Exclusion Criteria:

* Do not have a medical condition that prevents you from exercise (e.g. heart attack in the past year, heart disease, irregular heartbeat, etc.)
* Do not have history of eye injury or neurological impairment
* Do not have an orthopaedic limitation
* Are not pregnant

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Reaction Time | 30 minutes
  Time in milliseconds to target
Accuracy | 30 minutes
  Directional errors

OTHER OUTCOMES:
Heart Rate | 10 minutes
  Heart rate measured in beats per minute with a Polar Heart Rate Monitor as a manipulation check

CONTACTS AND LOCATIONS:
Overall Officials: Harry Prapavessis, Ph.D, Principal Investigator — Western University
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No